CLINICAL TRIAL: NCT01592305
Title: A Study to Evaluate the Potential Drug-Drug Interaction Between Danoprevir When Coadministered With Low-Dose Ritonavir and Tenofovir Disoproxil Fumarate or Atazanavir in Healthy Adult Volunteers
Brief Title: A Study of Drug-Drug Interaction Between Danoprevir Coadministered With Low-Dose Ritonavir and Tenofovir Disoproxil Fumarate or Atazanavir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None
Other Study IDs: NP28104
Record Dates: First submitted 2012-04-24; First posted 2012-05-07 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Atazanavir Sulfate; danoprevir; Ritonavir; Tenofovir

ARMS (3):
- S1 P1 TDF + DNV/r (Experimental)
  Interventions: Drug: danoprevir; Drug: ritonavir; Drug: tenofovir disoproxil fumarate
- S1/S2 P2 DNV/r + ATZ (Experimental)
  Interventions: Drug: atazanavir; Drug: danoprevir; Drug: ritonavir
- S2 P1 ATZ/r (Experimental)
  Interventions: Drug: atazanavir; Drug: ritonavir

INTERVENTIONS:
Drug: atazanavir — multiple oral doses
  Arms: S1/S2 P2 DNV/r + ATZ; S2 P1 ATZ/r
Drug: danoprevir — multiple oral doses
  Arms: S1 P1 TDF + DNV/r; S1/S2 P2 DNV/r + ATZ
Drug: ritonavir — multiple oral doses
Drug: tenofovir disoproxil fumarate — single oral doses
  Arms: S1 P1 TDF + DNV/r

SUMMARY:
This randomized, open-label, multiple-treatment multiple-dose, 2-period, 2-sequence study will evaluate potential drug-drug interactions between danoprevir (DNV) when coadministered with low-dose ritonavir (r) and tenofovir disoproxil fumarate (TDF) or atazanavir (ATZ) in healthy volunteers. Subjects will be randomized to receive in Period 1 either single oral doses of TDF and multiple oral doses of DNV/r or multiple oral doses of ATZ/r. In Period 2, all subjects will receive multiple oral doses of DNV/r plus ATZ. Anticipated time on study treatment is up to 20 days.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers, 18 to 55 years of age, inclusive
* Body weight >/= 55 kg
* Body mass index (BMI) 18.0 - 32.0 kg/m2
* Healthy non-smoking subjects. Healthy status will be defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history and a complete physical examination
* Medical history without major recent or ongoing pathology
* Females of childbearing potential and males and their female partners of childbearing potential must agree to use 2 forms of contraception, 1 of which must be a barrier method, during the study and for 90 days after the last drug administration

Exclusion Criteria:

* Pregnant or lactating women or males with female partners who are pregnant or lactating
* Any history of clinically significant disease or condition
* Positive for drugs of abuse at screening or prior to admission to the clinical site
* Positive for hepatitis B, hepatitis C or HIV infection
* Current smokers or subjects who have discontinued smoking less than 6 months prior to first dose of study medication
* Use of hormonal contraceptives (e.g. birth control pill, patches, or injectable, implantable devices) within 30 days before the first dose of study medication
* Use of an investigational drug or device within 30 days of the first dose of study medication (6 months for biologic therapies) or 5 half-lives of the investigational drug, whichever is longer
* History of drug-related allergy reaction
* History (within 3 months of screening) of alcohol consumption exceeding 2 standard drinks per day on average

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of tenofovir disoproxil fumarate and atazanavir when coadministered with danoprevir/ritonavir: Area under the concentration-time curve (AUC) | Pre-dose, and up to 48 hours post-dose Days 1, 8, 11, 16, 20
Pharmacokinetics of danoprevir and ritonavir when coadministered with tenofovir disoproxil fumarate and atazanavir: Area under the concentration-time curve (AUC) | Pre-dose, and up to 24 hours post-dose Days 10, 11, 16, 20

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | approximately 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Lenexa, Kansas, United States